CLINICAL TRIAL: NCT04991103
Title: Minimal Residual Disease Response-adapted Deferral of Transplant in Dysproteinemia - MILESTONE Trial
Brief Title: Minimal Residual Disease Response-adapted Deferral of Transplant in Dysproteinemia (MILESTONE)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Susan Bal, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300007387
Record Dates: First submitted 2021-07-27; First posted 2021-08-05 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma; Amyloidosis
Keywords: Minimal residual disease; Autologous stem cell transplantation
MeSH Terms: conditions — Multiple Myeloma; Amyloidosis; Neoplasm, Residual | interventions — daratumumab; Bortezomib; Lenalidomide; Dexamethasone; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: All patients with start with 6 cycles of quadruplet induction (Cohort A: daratumumab, lenalidomide, bortezomib and dexamethasone; Cohort B: daratumumab, cyclophosphamide, bortezomib and dexamethasone) and then depending of their response will receive additional consolidation/maintenance therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Daratumumab, Bortezomib, Dexamethasone with Lenalidomide/Cyclophosphamide (Experimental): Quadruplet therapy in the treatment of newly diagnosed myeloma and AL amyloidosis
  Interventions: Drug: DaraVRD/DaraVCD

INTERVENTIONS:
Drug: DaraVRD/DaraVCD — Patients in Cohort A with newly diagnosed multiple myeloma will receive six cycles of combination quadruplet therapy (DaraVRD).
  Six 28-day induction cycles of oral lenalidomide (25 mg daily on days 1-21), subcutaneous bortezomib (1.3 mg/m2 on days 1, 8, 15, 22), subcutaneous daratumumab (1800 mg on days 1, 8, 15, 22 of cycles 1-2 and days 1, 15 for cycles 3-6), and oral dexamethasone (40 mg on days 1, 8, 15, and 22).
  Patients in Cohort B with newly diagnosed amyloidosis will receive six cycles of combination quadruplet therapy (DaraVCD).
  Six 28-day induction cycles of IV cyclophosphamide (300 mg/m2 on days 1, 8, 15, 22), subcutaneous bortezomib (1.3 mg/m2 on days 1, 8, 15, 22), subcutaneous daratumumab (1800 mg on days 1, 8, 15, 22 of cycles 1-2 and days 1, 15 for cycles 3-6), and oral dexamethasone (40 mg on days 1, 8, 15, and 22).
  Other Names: daratumumab; bortezomib; lenalidomide; dexamethasone; cyclophosphamide

SUMMARY:
This is a phase II interventional study evaluating the use of minimal residual disease by next generation sequencing to defer autologous hematopoietic stem cell transplantation (AHCT) in patients with newly diagnosed multiple myeloma (cohort A) and amyloidosis (cohort B).

DETAILED DESCRIPTION:
While AHCT is an important treatment strategy for patients with plasma cell disorders, from a safety standpoint, AHCT is associated with both acute toxicities that reduce quality of life and long-term toxicities that may limit life expectancy for some patients. Additionally its benefit in patients without evidence of minimal residual disease (MRD) is unknown.

We propose to examine MRD response as a strategy to defer AHCT in a systematic manner.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years with no upper age limit with a diagnosis of newly diagnosed multiple myeloma with indication for initiation of therapy with Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* No prior therapy except for dexamethasone (up to 160 mg) and/or bortezomib (up to 5.2 mg/m2 ) and/or cyclophosphamide up to 1000 mg/m2 administered for management of acute manifestations of multiple myeloma (hypercalcemia, renal impairment, pain) for no longer than 4 weeks prior to enrollment (pre induction). If subject received any prior therapy, pretreatment parameters necessary for disease characterization and response assessment must be available.
* Measurable disease meeting at least one of the following criteria (at screening or prior to pre induction): 1) Serum monoclonal (M) protein ≥1.0 g/dl 2) ≥ 200 mg of M protein/24h in the urine 3) Serum free light chain ≥10 mg/dL and abnormal kappa to lambda ratio.
* Life expectancy ≥ 12 months.
* Adequate organ function - Hepatic function, with serum Alanine Aminotransferase ≤ 2.5 times the upper limit of normal and serum direct bilirubin ≤ 2 mg/dL (34 µmol/L) within 21 days prior to initiation of therapy. Creatinine clearance (CrCl) ≥ 40 mL/minute within 21 days prior to start of therapy.
* Females of childbearing potential (FCBP) must agree to ongoing pregnancy testing and to practice contraception during treatment and for 30 days after the last dose of bortezomib. Male subjects must agree to practice contraception and refrain from donating sperm during treatment and for 90 days after the last dose of bortezomib.
* All subjects must agree to comply with and be enrolled in Revlimid Risk Evaluation and Mitigation Strategy (REMS) program.
* Meet institutional criteria for autologous hematopoietic cell transplantation according to investigator's assessment.
* At least 30% ethnic/racial minorities will be included. If necessary, accrual will be held of non-ethnic minority patients while continuing for ethnic minorities in order to ensure at least 30% representation.

Exclusion Criteria:

* Diagnosis of POEMS (Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal protein, Skin changes), Waldenstrom's macroglobulinemia.
* Major surgery, radiotherapy or infection requiring therapy within 14 days of starting treatment.
* Pregnant or lactating females.
* Patients with uncontrolled human immunodeficiency virus, hepatitis B, hepatitis C. Patients may be eligible with Viral load is undetectable.
* Unstable angina or myocardial infarction within 4 months prior to registration, New York heart association Class II, III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker.
* Cerebrovascular disease manifested as prior stroke at any time or transient ischemic attack in the 12 months prior to initiation of therapy.
* Non hematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or localized thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas.
* Significant neuropathy (Grades 3-4, or Grade 2 with pain) within 21 days prior to registration.
* Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-08-27 (Estimated)

PRIMARY OUTCOMES:
Number of patients who are able to attain MRD<10-5 by next generation sequencing after 6 cycles of Dara-VRD and defer AHCT. | Baseline through 6 months
  To determine the feasibility of utilizing post-induction MRD to inform transplant utilization.

SECONDARY OUTCOMES:
Number of patients who was MRD>10-5 that undergo AHCT and attain MRD<10-5. | Baseline through 10 months
  To determine the frequency of conversion from MRD (+) to MRD (-) status with auto-HCT.
Progression free survival | Baseline through 7 years
  To determine the progression free survival (PFS)
Overall survival | Baseline through 7 years
  To determine the frequency of overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Bal, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
To be determined.